CLINICAL TRIAL: NCT04947514
Title: Use of TRanEXamic Acid in Reduction Mammoplasty (TREX-ARM): a Double-blinded Randomized Controlled Trial
Brief Title: Use of Tranexamic Acid in Reduction Mammoplasty
Acronym: TREX-ARM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: The Plastic Surgery Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-13090
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Results first posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Hematoma Postoperative; Venous Thromboembolism
Keywords: breast reduction mammoplasty; hematoma; tranexamic acid
MeSH Terms: conditions — Venous Thromboembolism; Hematoma | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Each patient undergoing routine bilateral breast reduction randomized to receive the study drug in either the right or left breast
Who Masked: Participant, Care Provider
Masking Description: The patient and the surgical team will be blinded to which breast has received the study drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Side (Right or Left) (Other): Each patient undergoing routine bilateral breast reduction will be randomized to receive the study drug (topical tranexamic acid) either to the right or left breast at the conclusion of the operation, prior to closure of the incisions. The other breast will receive topical saline.
  Interventions: Drug: Tranexamic acid
- Non-Treatment Side (Right or Left) (Other): Each patient undergoing routine bilateral breast reduction will be randomized to receive the study drug (topical tranexamic acid) either to the right or left breast at the conclusion of the operation, prior to closure of the incisions. The other breast will receive topical saline.
  Interventions: Other: Placebo (topical saline)

INTERVENTIONS:
Drug: Tranexamic acid — Topical tranexamic acid (1000mg) will be administered to the raw surface of the breast prior to closure of the incisions.
  Other Names: Cyklokapron
  Arms: Treatment Side (Right or Left)
Other: Placebo (topical saline) — The untreated breast will receive topical saline.
  Arms: Non-Treatment Side (Right or Left)

SUMMARY:
Breast reduction mammoplasty (BRM) is among the most commonly performed procedures in plastic surgery. However, postoperative hematoma is one of the most common complications following BRM. Hematoma-related complications include unplanned surgery, need for blood transfusion, wound healing issues, and unfavorable surgical outcomes.

Tranexamic acid has emerged in the literature as a promising agent that reduces perioperative blood loss and need for transfusion. However, despite its consistently reported efficacy, low cost, and favorable safety profile, tranexamic acid remains underutilized in plastic surgery.

The investigators propose a prospective, double-blinded randomized controlled study of the efficacy of tranexamic acid in reducing hematoma development in patients undergoing reduction mammoplasty. The investigators hope to contribute to the growing body of literature supporting tranexamic acid to reduce unwanted surgical bleeding.

DETAILED DESCRIPTION:
Prevention of perioperative blood loss is a chief consideration in plastic surgery. Breast reduction mammoplasty (BRM) is one of the most commonly performed procedures in plastic surgery, with over 100,000 performed in the United States in 2019 alone. Postoperative hematomas are among the most frequent complications following BRM, with a reported incidence between 0.3-7% in the literature. Many of these hematomas require blood transfusions and/or urgent surgical evacuation to avoid the consequent wound healing issues arising from increased tension on the closure.

Tranexamic acid (TXA) has emerged in the literature as a promising agent that reduces perioperative blood loss and need for transfusion. TXA is an antifibrinolytic agent that acts by stabilizing clot formation, and may be administered intravenously, orally, or topically. Topical administration of TXA has been shown to be as efficacious as intravenous dosing, though with substantially less systemic absorption. Multiple randomized controlled trials have demonstrated that TXA significantly reduces intraoperative bleeding and need for subsequent blood transfusion, without an increased risk of thromboembolic events. Moreover, TXA has been shown to be cost-effective in the surgical setting, not only by reducing direct hospital costs (drug and blood products), but also by decreasing subsequent costs by shortening length of stay and lowering the incidence of complications. However, the use of TXA in plastic surgery has not been well described.

The investigators propose a prospective, double-blinded randomized controlled study of the efficacy of TXA in patients undergoing BRM. The primary outcome variable will be the rate of hematoma development. The secondary outcome variables will be the incidence of blood transfusion and the incidence of thromboembolic events. The investigators will also collect a broad range of preoperative variables, surgical details, and other characteristics that may impact the perioperative bleeding risk. All patients eligible for reduction mammoplasty between July 1, 2021 and June 30, 2022 will be included in this study. The investigators hypothesize that use of TXA will decrease total perioperative blood loss, hematoma formation, and transfusion rates following reduction mammoplasty without increasing the incidence of thromboembolic events. Better understanding of the effect of TXA in reduction mammoplasty may be of great utility to the field of plastic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18
* Undergoing bilateral reduction mammoplasty at the Hutchinson Metro Center of Montefiore Medical Center, Bronx, New York

Exclusion Criteria:

* Oncologic breast reduction
* Unilateral breast reduction
* History of thromboembolic disease
* History of bleeding diatheses
* History of stroke
* History of seizure disorder
* Currently pregnant
* Severe comorbidity (defined as American Society of Anesthesiologists (ASA) fitness grade IV or above)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study population is patients undergoing breast reduction; typically, cisgender females elect to undergo breast reduction.
Enrollment: 98 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Ricci, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center Hutchinson Metro Center Campus, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaoutzanis C, Winocour J, Gupta V, Ganesh Kumar N, Sarosiek K, Wormer B, Tokin C, Grotting JC, Higdon KK. Incidence and Risk Factors for Major Hematomas in Aesthetic Surgery: Analysis of 129,007 Patients. Aesthet Surg J. 2017 Oct 16;37(10):1175-1185. doi: 10.1093/asj/sjx062. PMID 28398469
- [Background] Brown S, Yao A, Taub PJ. Antifibrinolytic Agents in Plastic Surgery: Current Practices and Future Directions. Plast Reconstr Surg. 2018 Jun;141(6):937e-949e. doi: 10.1097/PRS.0000000000004421. PMID 29794717
- [Background] Dadure C, Sauter M, Bringuier S, Bigorre M, Raux O, Rochette A, Canaud N, Capdevila X. Intraoperative tranexamic acid reduces blood transfusion in children undergoing craniosynostosis surgery: a randomized double-blind study. Anesthesiology. 2011 Apr;114(4):856-61. doi: 10.1097/ALN.0b013e318210f9e3. PMID 21358317
- [Background] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, Fergusson DA, Ker K. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2011 Jan 19;(1):CD001886. doi: 10.1002/14651858.CD001886.pub3. PMID 21249650
- [Background] Guerriero C, Cairns J, Perel P, Shakur H, Roberts I; CRASH 2 trial collaborators. Cost-effectiveness analysis of administering tranexamic acid to bleeding trauma patients using evidence from the CRASH-2 trial. PLoS One. 2011 May 3;6(5):e18987. doi: 10.1371/journal.pone.0018987. PMID 21559279
- [Background] Rohrich RJ, Cho MJ. The Role of Tranexamic Acid in Plastic Surgery: Review and Technical Considerations. Plast Reconstr Surg. 2018 Feb;141(2):507-515. doi: 10.1097/PRS.0000000000003926. PMID 28938364
- [Background] Weissler JM, Banuelos J, Jacobson SR, Manrique OJ, Nguyen MT, Harless CA, Tran NV, Martinez-Jorge J. Intravenous Tranexamic Acid in Implant-Based Breast Reconstruction Safely Reduces Hematoma without Thromboembolic Events. Plast Reconstr Surg. 2020 Aug;146(2):238-245. doi: 10.1097/PRS.0000000000006967. PMID 32740567
- [Background] Ausen K, Fossmark R, Spigset O, Pleym H. Randomized clinical trial of topical tranexamic acid after reduction mammoplasty. Br J Surg. 2015 Oct;102(11):1348-53. doi: 10.1002/bjs.9878. PMID 26349843
- [Background] Rubio GA, Zoghbi Y, Karcutskie CA, Thaller SR. Incidence and risk factors for venous thromboembolism in bilateral breast reduction surgery: An analysis of the National Surgical Quality Improvement Program. J Plast Reconstr Aesthet Surg. 2017 Nov;70(11):1514-1519. doi: 10.1016/j.bjps.2017.05.050. Epub 2017 Jun 2. PMID 28655514
- [Background] Xie J, Hu Q, Huang Q, Ma J, Lei Y, Pei F. Comparison of intravenous versus topical tranexamic acid in primary total hip and knee arthroplasty: An updated meta-analysis. Thromb Res. 2017 May;153:28-36. doi: 10.1016/j.thromres.2017.03.009. Epub 2017 Mar 10. PMID 28319822

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients undergoing bilateral reduction mammoplasty were enrolled in this study. One breast was randomized to receive the treatment, the other received a placebo; therefore, there were 98 patients enrolled and 196 "treated" breasts.
Units Other Than Participants: Breasts
Groups:
- Treatment Side (Tranexamic Acid) or Placebo Side (Topical Saline): Each patient undergoing routine bilateral breast reduction was randomized to receive the study drug (topical tranexamic acid) either to the right or left breast at the conclusion of the operation, prior to closure of the incisions. The other breast received topical saline.
  Treatment: Topical tranexamic acid (1000mg) will be administered to the raw surface of the breast prior to closure of the incisions.
  OR
  Placebo (topical saline): The untreated breast will receive topical saline.
Period: Overall Study
Arm/Group | Treatment Side (Tranexamic Acid) or Placebo Side (Topical Saline)
Started | 98; 196 Breasts
Completed | 98; 196 Breasts
Not Completed | 0; 0 Breasts

BASELINE CHARACTERISTICS:
Units Other Than Participants: Breasts
Arm/Group | Treatment Side (Tranexamic Acid) or Placebo Side (Topical Saline)
Number analyzed (Participants) | 98
Number analyzed (Breasts) | 196
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 98
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.14 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 3
  More than one race | 57
  Unknown or Not Reported | 20
Region of Enrollment [Number; unit: participants]
  United States | 98

OUTCOME MEASURES:

1. Primary Outcome: Number of Breasts With Development of Hematoma
Description: The number of breasts with clinically significant hematoma (collection of blood under the skin) requiring either conservative management or operative washout was determined.
Time Frame: Up to 30 days
Population: One of the two breasts was randomized to receive the study drug, the other breast was randomized to receive saline. As all participants had a bilateral operation performed, there were 196 analyzed units for 98 participants.
Measure: Number; unit: breasts
Units Other Than Participants: Breast
Groups:
- Placebo Side (Right or Left): Each patient undergoing routine bilateral breast reduction will be randomized to receive the study drug (topical tranexamic acid) either to the right or left breast at the conclusion of the operation, prior to closure of the incisions. The other breast will receive topical saline.
  Placebo (topical saline): The untreated breast will receive topical saline.
Arm/Group | Treatment Side (Right or Left) | Placebo Side (Right or Left)
Number analyzed (Participants) | 98 | 98
Number analyzed (Breast) | 98 | 98
breasts | 2 | 1

2. Secondary Outcome: Number of Participants Requiring a Blood Transfusion
Description: The number of participants requiring blood transfusion was based on the postoperative decline in hematocrit level
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Side (Right or Left) | Placebo Side (Right or Left)
Number analyzed (Participants) | 98 | 98
Participants | 0 | 0

3. Secondary Outcome: Number of Participants With Deep Vein Thrombosis/Venous Thromboembolism
Description: Incidence of clinically significant deep vein thrombosis or pulmonary embolism detected on imaging (ultrasound or CT scan)
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Side (Right or Left) | Placebo Side (Right or Left)
Number analyzed (Participants) | 98 | 98
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 1 week postoperatively
Arm/Group | Treatment Side (Right or Left) | Placebo Side (Right or Left)
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/98
Other Adverse Events (participants affected / at risk) | 0/98 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT04947514/Prot_SAP_000.pdf